CLINICAL TRIAL: NCT03256669
Title: Umblical Incision for Neonatal Surgey; is it Suitable
Brief Title: Umblical Incision for Neonatal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Abdelmalek, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1a765
Record Dates: First submitted 2017-07-29; First posted 2017-08-22 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Neonatal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- umbilical incision (Experimental): neonates undergone surgery by umbilical incision
  Interventions: Procedure: umbilical incision

INTERVENTIONS:
Procedure: umbilical incision — exploration through umbilical incision

SUMMARY:
Abdominal exploration leave an ugly scar that live with the baby forever, laparoscopy can solve the problem to some extent by making a smaller scar but takes more time and need special surgical skills. Umbilical incision can combine the advantage of open and laparoscopy and avoid the drawbacks of both.

DETAILED DESCRIPTION:
six cases were subjected to the study 2 cases have duodenal atresia, one case has annular pancreas, one case has jujenal atresia chritmas tree, one case has jujenal web and a case of malrotation. all of them had made exploration by the umbilical incision, and no drains had been used.

ELIGIBILITY:
Inclusion Criteria:

* neonate diagnosed radiologically

Exclusion Criteria:

* unclear diagnosis

Ages: 20 Hours to 20 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
operative time | 2 hours
  how long the peration does take

SECONDARY OUTCOMES:
cosmotic appearance | 2 weeks
  shape of the wound

OTHER OUTCOMES:
result | 1 week
  surgical result successful or not

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No